CLINICAL TRIAL: NCT05299242
Title: Anti-TNF (Adalimumab) Injection for the Treatment of Adults With Frozen Shoulder During the Pain-predominant Phase: a Multi-centre, Randomised, Double Blind, Parallel Group, Feasibility Study
Brief Title: The Anti-Freaze-F Study- "Anti-TNF for Treatment of Frozen Shoulder - a Feasibility Study"
Acronym: Anti-FreazeF
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); 180 Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: 15701
Record Dates: First submitted 2022-02-17; First posted 2022-03-28 (Actual); Results first posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2022-11

CONDITIONS: Frozen Shoulder
Keywords: Adhesive capsulitis
MeSH Terms: conditions — Bursitis | interventions — Adalimumab

STUDY DESIGN:
Intervention Model Description: Participants will be randomised to either receive Adalimumab or Placebo.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant will be blinded along with the assessor and other site staff. The injector and pharmacy will not be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): Participants will receive 2 injections of adalimumab. First injection: 160mg in 3.2ml Second injection approximately 2-3 weeks later 80mg in 1.6ml
  Interventions: Drug: Adalimumab Injection
- Arm B (Placebo Comparator): Participants will receive 2 injections of placebo First injection: 3.2ml Second injection approximately 2-3 weeks later 1.6ml
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Adalimumab Injection — 40mg in 0.8ml preparation in vials from Fresenius Kabi Ltd
  Arms: Arm A
Drug: Placebo — Saline [0.9% NaCl]
  Arms: Arm B

SUMMARY:
Frozen shoulder is a common condition affecting approximately 9% of people aged 25-64 years. During the early phase the pain is usually unbearable and the later restriction in movement is severely limiting. It occurs when the flexible tissue (capsule) that surrounds the shoulder joint becomes inflamed, thickened and tight. The pain can be very severe and lasts 3-9 months, followed by a 4-12 month period of increasing stiffness, after which the condition usually improves. Frozen shoulder often affects a person's ability to sleep, carry out everyday activities, and work. Current treatments include rest, painkillers, anti-inflammatories, physiotherapy and steroid injections. If stiffness persists, surgery is sometimes recommended. However, there is no evidence that any of these treatments lead to significant benefit in the long term, with many being ineffective. The aim of this study is to find out if it is possible to run a larger trial to test whether an injection of adalimumab can reduce pain and prevent the disease from getting worse, if given during the early painful phase of frozen shoulder. The investigators need to conduct this smaller study first to be sure it's possible to identify and treat people with early stage frozen shoulder, before they conduct a much larger trial to find out if this treatment works.

In this study the investigators will include 84 adults from 5 sites with painful early stage frozen shoulder who have not yet received treatment. People will be randomised to receive either an injection of the drug adalimumab or a dummy injection of saline (placebo) directly into the shoulder joint, both guided by ultrasound. All participants will also receive standardized advice on how to manage their shoulder pain. The investigators will assess participants before treatment and three months later. Adalimumab has been used very successfully to treat other inflammatory diseases such as rheumatoid arthritis. This study has been funded by the NIHR RfPB programme and 180 Life Sciences.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 years and above.
2. With a new episode of shoulder pain attributable to pain-predominant stage of frozen shoulder (i.e. within approximately 3 months of onset of symptoms) diagnosed using criteria set out in the BESS guidelines (33) (Appendix 1);
3. Who are not being considered for surgery;
4. Able to understand spoken and written English;
5. Willing and able to give informed consent for trial participation and comply with all study requirements and time line;
6. Willing to allow his or her General Practitioner be notified of participation in the trial.
7. If female and of child-bearing potential OR if male and their partner is of child-bearing potential - willing to use effective contraception throughout the treatment period and for 5 months after the last injection.-

Exclusion Criteria:

1. Those with frozen shoulder secondary to significant shoulder trauma (e.g., dislocation, fracture or full thickness tear requiring surgery) or other causes (e.g. recent breast cancer surgery or radiotherapy);
2. Those with a neurological disease affecting the shoulder;
3. Those with bilateral concurrent frozen shoulder;
4. Those with other shoulder disorders (e.g., inflammatory arthritis, rotator cuff disorders, glenohumeral joint instability) or with red flags consistent with the criteria set out in the BESS guidelines (33);
5. Those who have received corticosteroid injection for shoulder pain in the last 12 weeks to either shoulder;
6. Those currently taking any anti-TNF drug;
7. Those being treated with coumarin anticoagulants, such as warfarin;
8. Those who have participated in another research study involving an investigational medicinal product in the past 12 weeks;
9. Those with significant renal or hepatic impairment;
10. Those with contra-indications to anti-TNF injection:

10.1 Known allergy to any anti-TNF agent or any of the excipients; 10.2 Known Active tuberculosis (TB) or history of TB. 10.3 Known Active infection (chronic or localised) or known history of recurring infections or condition which may predispose patients to infection, including the use of concomitant immunosuppressive medications; 10.4 Known Moderate to severe heart failure (NYHA class III/IV); 10.5 Those known to have HIV, Hepatitis B or C; 10.6 Those at risk of Hepatitis B infection; 10.7 Those diagnosed with Multiple Sclerosis (MS) or other central or peripheral nervous system demyelinating disorders; 10.8 Those who have ever been diagnosed with cancer, except basal cell carcinoma (BCC); 10.9 Those requiring live vaccination prior to within 12 weeks after of the last trial injection or within the 4 weeks prior to randomisation; 10.10 Those taking biologic DMARDS; 10.11 Any other significant disease or disorder which, in the opinion of the Investigator, may either put the participants at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 9 (Actual)
Dates: Start 2022-07-21 (Actual); Primary Completion 2023-05-09 (Actual); Study Completion 2023-06-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jagdeep Nanchahal, Principal Investigator — University of Oxford
Locations (4):
- United Kingdom (4):
  - Good Hope Hospital, Sutton Coldfield, Birmingham
  - Conquest Hospital, Saint Leonards-on-Sea, Hastings
  - Grantham & District Hospital, United Lincolnshire Hospitals, Grantham, Lincolnshire
  - Sandwell General Hospital, West Bromwich, West Midlands

IPD SHARING:
Plan to Share IPD: Yes
Summary results data will be available on the trial registration database within 12 months of the end of the trial. Requests for data (anonymised participant data) will only be provided at the end of the trial to external researchers who provide a methodologically sound proposal to the trial team aff@kennedy.ox.ac.uk (will be required to sign a data sharing access agreement with the Sponsor) and in accordance with the NIHR guidance. Participant consent for this is included in the informed consent form for the study
Supporting Information: Study Protocol
Access Criteria: Available on request

REFERENCES:
- [Background] Hopewell S, Kenealy N, Knight R, Rangan A, Dutton S, Srikesavan C, Feldmann M, Lamb S, Nanchahal J. Anti-TNF (adalimumab) injection for the treatment of adults with frozen shoulder during the pain predominant stage protocol for a multi-centre, randomised, double blind, parallel group, feasibility trial. NIHR Open Res. 2023 Apr 24;2:28. doi: 10.3310/nihropenres.13275.2. eCollection 2022. PMID 37881307
- [Derived] Hopewell S, Srikesavan C, Evans A, Er F, Rangan A, Preece J, Francis A, Massa MS, Feldmann M, Lamb S, Nanchahal J. Anti-TNF (adalimumab) injection for the treatment of pain-predominant early-stage frozen shoulder: the Anti-Freaze-Feasibility randomised controlled trial. BMJ Open. 2024 May 1;14(5):e078273. doi: 10.1136/bmjopen-2023-078273. PMID 38692727
- See also: Results Paper (BMJ Open) — http://bmjopen.bmj.com/content/14/5/e078273.long
- See also: Protocol Paper (NIHR Open Research) — http://openresearch.nihr.ac.uk/articles/2-28

RESULTS

PARTICIPANT FLOW:
Groups:
- Adalimumab: Participants received 2 injections of adalimumab. First injection: 160mg in 3.2ml. Second injection approximately 2-3 weeks later: 80mg in 1.6ml.
  Adalimumab Injection: 40mg in 0.8ml preparation in vials from Fresenius Kabi Ltd.
- Placebo: Participants received 2 injections of placebo. First injection: 3.2ml. Second injection approximately 2-3 weeks later: 1.6ml.
  Placebo: Saline [0.9% NaCl]
Period: Overall Study
Arm/Group | Adalimumab | Placebo
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Adalimumab | Placebo | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.5 (5.9) | 52.8 (5.0) | 54.9 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 2 | 3
  Male | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White British | 4 | 5 | 9
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 4 | 5 | 9
Handedness [Count of Participants; unit: Participants]
  Left | 2 | 1 | 3
  Right | 2 | 4 | 6
Duration of symptoms [Mean (Standard Deviation); unit: weeks] | 19.5 (13.1) | 12.2 (2.3) | 15.4 (9.0)
Smoking status [Count of Participants; unit: Participants]
  Never smoked | 4 | 3 | 7
  Former smoker | 0 | 2 | 2
Dupuytren's disease [Count of Participants; unit: Participants]
  No | 4 | 4 | 8
  Yes | 0 | 1 | 1
Diabetes [Count of Participants; unit: Participants]
  Type 1 | 0 | 1 | 1
  Type 2 | 1 | 2 | 3
  No | 3 | 2 | 5
If ever smoked, number of cigarettes/day [Mean (Standard Deviation); unit: cigarettes per day] — Population: There were no participants in the Adalimumab group who were smokers, therefore the number of cigarettes smoked per day could not be collected for this group.
  cigarettes per day
    number analyzed (Participants) | 0 | 5 | 5
    (all) |  | 12 (11.3) | 12 (11.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Eligible With Pain Predominant Frozen Shoulder
Description: Ability to screen and identify potential participants with pain-predominant early stage frozen shoulder (i.e. within approximately 3 months of onset of symptoms).
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Groups:
- All Screened Participants: All participants who were screened for pain predominant frozen shoulder.
Arm/Group | All Screened Participants
Number analyzed (Participants) | 156
Participants | 39

2. Primary Outcome: Number of Participants Consenting to be Included in the Trial
Description: Willingness of eligible participants to consent and be randomised to intervention.
Time Frame: 3 Months
Measure: Count of Participants; unit: Participants
Groups:
- Eligible Participants: All participants deemed eligible for the trial after screening.
Arm/Group | Eligible Participants
Number analyzed (Participants) | 39
Participants | 9

3. Primary Outcome: Time From Randomisation to First Injection
Description: Practicalities of delivering the intervention, including time to first injection (within 2 weeks of randomisation).
Time Frame: 2 weeks
Population: All participants received their treatment as allocated and in line with the trial protocol. One participant in the adalimumab group received their injection 18 days post- randomisation as they were not available until then.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Adalimumab | Placebo
Number analyzed (Participants) | 4 | 5
days | 12.3 (4.8) | 7.2 (4.1)

4. Primary Outcome: Time From First Injection to Second Injection
Description: Practicalities of delivering the intervention, including time between first injection and second injection (within 4-6 weeks of randomisation).
Time Frame: 6 weeks
Population: All participants received their treatment as allocated and in line with the trial protocol.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Adalimumab | Placebo
Number analyzed (Participants) | 4 | 5
days | 18.5 (3.3) | 20.8 (5.9)

5. Primary Outcome: Shoulder Pain and Disability Index (SPADI) Score
Description: Score ranges from 0 to 100, lower scores indicate better outcome.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adalimumab | Placebo
Number analyzed (Participants) | 4 | 5
score on a scale
  Baseline | 70.8 (16.6) | 55.4 (21.5)
  3 months | 40.1 (30.0) | 45.8 (25.3)

6. Secondary Outcome: Pain (Shoulder Pain And Disability Index, 5-item Subscale)
Description: Score ranges from 0 to 100, lower scores indicate better outcome.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adalimumab | Placebo
Number analyzed (Participants) | 4 | 5
score on a scale
  Baseline | 78.5 (18.4) | 63.2 (19.5)
  3 months | 41.5 (32.7) | 49.6 (27.3)

7. Secondary Outcome: Function (Shoulder Pain And Disability Index, 8-item Subscale)
Description: Score ranges from 0 to 100, lower scores indicate better outcome.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adalimumab | Placebo
Number analyzed (Participants) | 4 | 5
score on a scale
  Baseline | 63.1 (15.6) | 47.5 (25.7)
  3 months | 38.8 (30.3) | 42.0 (24.7)

8. Secondary Outcome: Fear Avoidance Belief Questionnaire
Description: Score ranges from 0 to 24, higher scores indicate better outcomes.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adalimumab | Placebo
Number analyzed (Participants) | 4 | 5
score on a scale
  Baseline | 17.3 (3.3) | 17.4 (3.6)
  3 months | 9.3 (6.2) | 12.8 (5.9)

9. Secondary Outcome: Pain Self Efficacy Questionnaire
Description: Score ranges from 0 to 12, higher scores indicate better outcomes.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adalimumab | Placebo
Number analyzed (Participants) | 4 | 5
score on a scale
  Baseline | 9 (3.6) | 9.2 (1.9)
  3 months | 10.5 (1.3) | 8.2 (2.8)

10. Secondary Outcome: Insomnia Severity Index
Description: Sleep disturbance measured using the Insomnia Severity Index, score ranges from 0 to 28, higher scores indicate worse outcomes.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adalimumab | Placebo
Number analyzed (Participants) | 4 | 5
score on a scale
  Baseline | 17.8 (5.0) | 17.6 (4.0)
  3 months | 9.8 (6.7) | 13.2 (7.6)

11. Secondary Outcome: Return to Desired Activities (RDA)
Description: Return to desired activities measured using an adapted version of the Disabilities of the Arm, Shoulder and Hand (QUICKDASH) questionnaire. Score ranges from 3 to 15, lower scores indicate better outcomes.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adalimumab | Placebo
Number analyzed (Participants) | 4 | 5
score on a scale
  Baseline | 9.0 (4.5) | 9.4 (2.7)
  3 month | 5.5 (3.8) | 8.4 (3.6)

12. Secondary Outcome: Global Impression of Change
Description: This was measured using the Likert scale. Score ranges from -5 (very much worse) to +5 (completely recovered) with a value of 0 suggesting no change. Higher scores indicate better outcomes.
Time Frame: 3 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Adalimumab | Placebo
Number analyzed (Participants) | 4 | 5
score on a scale | 2.3 (2.2) | 0.0 (3.0)

13. Secondary Outcome: Health Resource Use
Description: Consultation with primary and secondary care, additional physiotherapy, injection use, or alternative therapies for index shoulder
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Adalimumab | Placebo
Number analyzed (Participants) | 4 | 5
Participants
  Steroid injection (injection outside of the trial): Yes | 1 | 0
  Steroid injection (injection outside of the trial): No | 3 | 5
  NHS community-based services (physiotherapist): Yes | 1 | 0
  NHS community-based services (physiotherapist): No | 3 | 5
  Hospital as NHS outpatient (physiotheraphy department): Yes | 2 | 0
  Hospital as NHS outpatient (physiotheraphy department): No | 2 | 5
  Admitted as an inpatient: Yes | 0 | 0
  Admitted as an inpatient: No | 4 | 5
  Had surgery: Yes | 0 | 0
  Had surgery: No | 4 | 5

14. Secondary Outcome: Adverse Events Graded 3 or Above
Description: Any adverse event (graded 3 or above) that has resulted from the trial.
  The Common Terminology Criteria for Adverse Events (CTCAE) v5.0 was used to guide recording adverse events including grading of the event. Grade 3: Severe symptoms or medically significant but not life-threatening but may be disabling or limit self care in Activities of Daily Living. Grade 4: Life threatening consequences; urgent or emergent intervention needed. Grade 5: Death related to or due to adverse event.
Time Frame: Consent to 3 months follow-up
Measure: Number; unit: Adverse events graded 3 or above
Arm/Group | Adalimumab | Placebo
Number analyzed (Participants) | 4 | 5
Adverse events graded 3 or above | 0 | 0

15. Secondary Outcome: Shoulder Range of Movement
Description: Clinician assessed (goniometry measured) active shoulder flexion, extension, abduction, internal and external rotation. Range of flexion and abduction: 0-180 degrees. Range of extension, internal rotation and external rotation: 0-90 degrees.
Time Frame: Baseline and 3 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Adalimumab | Placebo
Number analyzed (Participants) | 4 | 5
degrees
  Baseline flexion | 71.3 (26.3) | 101.6 (24.7)
  3-month flexion | 112.5 (54.8) | 140.0 (25.7)
  Baseline extension | 26.3 (18.0) | 27.6 (9.5)
  3-month extension | 30.0 (8.2) | 40.6 (9.8)
  Baseline abduction | 50.0 (30.3) | 69.0 (26.6)
  3-month abduction | 105.0 (56.1) | 115.0 (42.7)
  Baseline internal rotation | 23.8 (18.9) | 40.2 (40.8)
  3-month internal rotation | 21.3 (17.0) | 41.0 (37.8)
  Baseline external rotation | 22.5 (8.7) | 15.0 (16.9)
  3-month external rotation | 28.8 (6.3) | 55.0 (16.2)

ADVERSE EVENTS:
Time Frame: From consent to 3 months follow-up.
Arm/Group | Adalimumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

LIMITATIONS AND CAVEATS:
This study demonstrated that current NHS musculoskeletal physiotherapy settings yielded only small numbers of participants, too few to make a trial viable. This was because many patients had passed the early stage of frozen shoulder or had already formulated a preference for treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/42/NCT05299242/Prot_SAP_000.pdf